CLINICAL TRIAL: NCT00219050
Title: An Eight-week, Randomized, Double-blind, Multi-center, Active-controlled, Parallel Group Study to Evaluate the Safety and Efficacy of an Aliskiren-based Regimen Compared to a Lisinopril-based Regimen in Patients With Uncomplicated Severe Hypertension
Brief Title: A Clinical Study to Compare the Safety and Efficacy of an Aliskiren-based Regimen With a Lisinopril Based Regimen in Patients With Severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2303
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
To compare the safety and efficacy of an aliskiren-based regimen to a lisinopril-based regimen in the treatment of severe hypertension

ELIGIBILITY:
Inclusion Criteria

* Patients with essential severe hypertension Exclusion Criteria
* History or evidence of a secondary form of hypertension
* History of hypertensive encephalopathy or cerebrovascular accident.
* Diabetic patients requiring insulin Other protocol-defined inclusion/exclusion criteria also apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2005-02; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Evaluate safety through adverse events and laboratory abnormalities after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in diastolic blood pressure after 8 weeks
Change from baseline in systolic blood pressure after 8 weeks
Change from baseline in standing systolic blood and diastolic pressure after 8 weeks
Diastolic blood pressure is less than 90 mmHg or reduction of 10 mmHg or greater from baseline after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Investigative Site, Berlin, Germany
- Investigative Site, Budapest, Hungary
- Investigative Site, Madrid, Spain
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Derived] Wang GM, Li LJ, Fan L, Xu M, Tang WL, Wright JM. Renin inhibitors versus angiotensin receptor blockers for primary hypertension. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD012570. doi: 10.1002/14651858.CD012570.pub2. PMID 40013543
- [Derived] Wang GM, Li LJ, Tang WL, Wright JM. Renin inhibitors versus angiotensin converting enzyme (ACE) inhibitors for primary hypertension. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD012569. doi: 10.1002/14651858.CD012569.pub2. PMID 33089502